CLINICAL TRIAL: NCT03349905
Title: A Randomized Trial of Deferred Versus Fresh Embryo Transfers in Infertile Women Undergoing IVF-ICSI
Brief Title: Deferred Versus Fresh Embryo Transfers
Acronym: DEFETOSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AOM160313
Record Dates: First submitted 2017-11-17; First posted 2017-11-22 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Infertility, Female
Keywords: Freeze all; IVF; deferred embryo transfer; endometriosis
MeSH Terms: conditions — Infertility, Female; Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fresh transfer (Active Comparator): Women randomized in the non experimental group will have:
  * Antagonist stimulation protocol
  * Ovarian triggering using a single injection of rhCG (Ovitrelle®; Serono, France)
  * All of their embryo kept in prolonged culture
  * A fresh single embryo transfer at blastocyst stage (on day 5 or 6 according to blastocyst stage)
  * Supernumerary blastocysts cryopreserved
  Interventions: Procedure: fresh transfer
- Deferred-frozen embryo transfer (Experimental): Women randomized in the experimental group will have:
  * Antagonist stimulation protocol
  * Ovarian triggering using a single injection of 0.2 mg of GnRH agonist triptorelin (Decapeptyl® Ipsen France)
  * All of their embryo cryopreserved at the blastocyst stage after prolonged embryo culture.
  * A frozen-thawed single embryo transfer at blastocyst stage, is planned 3-11 weeks after cryopreservation
  Interventions: Procedure: Deferred-frozen embryo transfer

INTERVENTIONS:
Procedure: fresh transfer — Women randomized in the non experimental group will have:
  * Antagonist stimulation protocol
  * Ovarian triggering using a single injection of rhCG (Ovitrelle®; Serono, France)
  * All of their embryo kept in prolonged culture
  * A fresh single embryo transfer at blastocyst stage (on day 5 or 6 according to blastocyst stage)
  * Supernumerary blastocysts cryopreserved
  Arms: Fresh transfer
Procedure: Deferred-frozen embryo transfer — Women randomized in the experimental group will have:
  * Antagonist stimulation protocol
  * Ovarian triggering using a single injection of 0.2 mg of GnRH agonist triptorelin (Decapeptyl® Ipsen France)
  * All of their embryo cryopreserved at the blastocyst stage after prolonged embryo culture.
  * A frozen-thawed single embryo transfer at blastocyst stage, is planned 3-11 weeks after cryopreservation
  Arms: Deferred-frozen embryo transfer

SUMMARY:
Controlled ovarian stimulation (COS) enhances the efficacy of ART (Assisted reproductive technology) by permitting multiple-oocyte yields, but also alters endometrial receptivity (ER) by an advancement of endometrial development which contributes to diminished pregnancy chances. Previous reports suggest that pregnancy rates are increased following deferred frozen embryo transfers. In addition as compared to fresh embryo transfers, frozen embryo transfers seem to be associated with less affected perinatal outcomes, in particular lower risk of preterm birth, small for gestational age and caesarean section. Unfortunately, most of the current evidence is based only on preliminary reports, needing further scientific evidence. Thus, whether differing embryo transfers could restore optimal ER leading to higher live birth rate (LBR) and better obstetrical outcomes as compared to fresh embryo transfers, is actually still under investigation.

DETAILED DESCRIPTION:
Controlled ovarian stimulation (COS) enhances the efficacy of ART (Assisted reproductive technology) by permitting multiple-oocyte yields, but also alters endometrial receptivity (ER) by an advancement of endometrial development which contributes to diminished pregnancy chances. Recently, technical improvements in vitrification make frozen embryo transfers (FETs) a safe and feasible alternative to fresh embryo transfer (Evans et al., 2014). In case of FET the absence of COS avoid the alteration of endometrial receptivity. Previous reports suggest that pregnancy rates are increased and perinatal outcomes are less affected following FET (Evans et al., 2014). In fact previous studies plead for increased risk of preterm birth, small for gestational age, caesarean section after fresh embryo transfer as compared to frozen embryo transfer (Maheshwari et al., 2012). Unfortunately, most of the current evidence is based only on preliminary reports, needing further scientific evidence. Thus, one of the main questions, in the management of infertile women, is to know whether differing embryo transfers could restore optimal endometrial receptivity leading to higher live birth rate (LBR) and better obstetrical outcomes as compared to fresh embryo transfer. This question is actually debated in the literature in many different reviews (Blockeel et al., 2016; Cedars, 2016; Engmann et al., 2016; Evans et al., 2014; Roque, 2015). However even if the scientific rationale is in favour of increased pregnancy rates after differed FET, compelling clinical evidence is still lacking and most of the current evidence is based on retrospective and uncontrolled studies. Currently the best evidence come from a very recent randomized control trial of fresh versus frozen embryo transfers in a specific population of polycystic ovary syndrome affected women (Chen et al., 2016). The authors failed to show any difference in pregnancy rate after fresh versus frozen embryo transfers but they found higher rate of miscarriages after fresh embryo transfers and in consequence a slight but significant decrease in live birth after fresh as compared to frozen embryo transfers (Chen et al., 2016). However whether these results, coming from a specific population of polycystic ovary syndrome affected women, may be generalizable is actually still unknown. Furthermore some evidence come from a meta-analysis, including 3 randomized studies. The conclusions of this meta-analysis are that IVF outcomes may be improved by performing FET compared with fresh embryo transfer probably through an improvement of endometrial receptivity (Roque et al., 2013). Nevertheless, this meta-analysis should be interpreted with caution. One of the included studies had been retracted from literature because of methodological problem (Aflatoonian et al., 2010). Therefore, this meta-analysis banking on a retracted study seems no more valid and therefore its conclusions remained uncertain. Even in absence of solid clinical studies and even in absence of valid recommendations, some authors conclude that IVF outcomes can be improved using the freeze-all policy with differed FET (Roque et al., 2015). In addition they recommend that further randomized clinical trials are needed to confirm the advantage of this strategy and determine the population for which it would be most beneficial. This last point seems crucial as ART procedures (IVF-ICSI) encompass a mixture of different fertility problem more or less sensible to the effects of COS on endometrial receptivity. Among the different causes of infertility, endometriosis is quite common and up to 20 % of women undergoing ART have associated endometriosis (Kawwass et al., 2015; Kuivasaari-Pirinen et al., 2012; Senapati et al., 2016). In addition endometriosis is characterized by impaired endometrial receptivity, contributing to the mechanisms by which endometriosis interfere with fecundity (de Ziegler et al., 2010). Estimated prevalence of endometriosis range from 2 to 10% of women of reproductive age, to 50% of infertile women (Eskenazi and Warner, 1997; Meuleman et al., 2009). Reverting to ART in case of endometriosis related infertility remain a solid option. However recent meta-analysis evocates decreased live birth rate in case of severe endometriosis as compared to disease free women (Hamdan et al., 2015). In addition endometriosis may be associated to adverse obstetrical outcomes (Leone Roberti Maggiore et al., 2016). Thus, given the existence of altered endometrial receptivity in endometriosis, and diminished ART outcomes, it is actually also debated whether deferring embryo transfers could restore optimal endometrial receptivity leading to higher live birth rate and reduced obstetrical risk in endometriosis affected women.

ELIGIBILITY:
Inclusion Criteria:

* Women [18 - 40[years of age (according to date of birth at time of informed consent) who are eligible for ovarian stimulation and ART treatment, including intracytoplasmic sperm injection (ICSI)
* Absence of anatomical abnormalities of the reproductive tract that would interfere with implantation or pregnancy
* Absence of any medical condition in which pregnancy is contraindicated
* Motile, ejaculatory sperm must be available (donated and/or cryopreserved sperm is allowed). Intracytoplasmic sperm injection (ICSI) will be allowed during this trial
* Body mass index 18 to 35 kg/m2, inclusive
* Able to understand the study
* Affiliation with a social security scheme
* Dated and signed inform consent

Exclusion Criteria:

* Altered ovarian reserve (Day3: FSH >12 UI/l; AMH<1,0 ng/ml; AFC<8)
* History or presence of tumours of the hypothalamus or pituitary gland
* Presence of non isolated uni- or bilateral hydrosalpinx
* Abnormal gynaecological bleeding of undetermined origin
* Contraindication to being pregnant and/or carrying a pregnancy to term
* Known infection with human immunodeficiency virus, active hepatitis B or C virus in the female or male partner
* History or presence of ovarian, uterine or mammary cancer
* Known allergy or hypersensitivity to human gonadotropin preparations or to compounds that are structurally similar to any of the other medications administered during the trial
* Substance abuse that would interfere with trial conduct, as determined by the investigator
* Use of testicular or epididymal sperm
* Pregnant patient, nursing patient
* Participation in another ART clinical trial within the past 30 days
* Women who have risk to develop severe ovarian hyperstimulation syndrome (OHSS) during controlled ovarian stimulation (COS) defined as ≥ 18 follicles measuring 10 - 14 mm on the day of triggering
* Women with less than 3 follicles ≥ 15 mm on the triggering day or the day before the triggering
* Women with premature progesterone elevation during COS ( ≥1.5 ng/ml)
* Women with uterine polyps diagnosed during COS
* Participation with another interventional study involving human subjects

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 237 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2022-01-19 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Live birth rates | ≥ 35 weeks of gestation after the first single blastocyst embryo transfer according to fresh or deferred-frozen transfer.
  The cut-off of 35 weeks postmenstrual age is to ensure the health and well being of the newborns babies.

SECONDARY OUTCOMES:
Miscarriage | ≥ 35 weeks of gestation after the first single blastocyst embryo transfer a
  Miscarriage is defined as an intrauterine clinical pregnancy that occurs before 20 completed weeks postmenstrual age (18 weeks post fertilization). Clinical pregnancy is defined as a pregnancy diagnosed by ultrasonographic visualization of one or more gestational sacs or definitive clinical signs of pregnancy. It includes ectopic pregnancy
Preterm birth | ≥ 35 weeks of gestation after the first single blastocyst embryo transfer a
  Preterm birth is defined as a live birth or stillbirth that takes place after at least 20 but before 37 completed weeks of postmenstrual age.
Preterm rupture of membranes | ≥ 35 weeks of gestation after the first single blastocyst embryo transfer a
  s defined as rupture of the foetal membranes occurring before labour and prior to 37 weeks of postmenstrual age.
Pre-eclampsia | ≥ 35 weeks of gestation after the first single blastocyst embryo transfer a
  is defined as gestational hypertension (Blood pressure ≥ 14 mm Hg systolic or ≥ 9 mm Hg diastolic, measured on two occasions at least four hours apart) associated with proteinuria ≥ 0.3 grams (300 mg) or more of protein in a 24-hour urine sample.
Placenta praevia | ≥ 35 weeks of gestation after the first single blastocyst embryo transfer a
  is defined by the presence of lower edge of the placenta < 50 mm behind the internal cervical os as diagnosed during the obstetrical ultrasound during the third trimester of the pregnancy. We also defined as placenta praevia when placenta partially or completely covers the internal cervical.
Live birth rates in Endometriosis related infertility | ≥ 35 weeks of gestation after the first single blastocyst embryo transfer a
  Analysis of live birth among women with endometriosis related infertility
Number of oocytes retrieved | ≥ 35 weeks of gestation after the first single blastocyst embryo transfer according to fresh or deferred-frozen transfer.
Number of MII oocytes | ≥ 35 weeks of gestation after the first single blastocyst embryo transfer according to fresh or deferred-frozen transfer.
Number of embryo | ≥ 35 weeks of gestation after the first single blastocyst embryo transfer according to fresh or deferred-frozen transfer.
Number of blastocyst | ≥ 35 weeks of gestation after the first single blastocyst embryo transfer according to fresh or deferred-frozen transfer.
Number of transferred blastocyst | ≥ 35 weeks of gestation after the first single blastocyst embryo transfer according to fresh or deferred-frozen transfer.
The cancellation rate | ≥ 35 weeks of gestation after the first single blastocyst embryo transfer according to fresh or deferred-frozen transfer.
The rate of started pregnancy | ≥ 35 weeks of gestation after the first single blastocyst embryo transfer according to fresh or deferred-frozen transfer.
The rate of pregnancy confirmed by the Echography (cardiac activity) | ≥ 35 weeks of gestation after the first single blastocyst embryo transfer according to fresh or deferred-frozen transfer.
Started pregnancy defined by a rate of HCG>100 | ≥ 35 weeks of gestation after the first single blastocyst embryo transfer according to fresh or deferred-frozen transfer.
Rate of multiple pregnancy | ≥ 35 weeks of gestation after the first single blastocyst embryo transfer according to fresh or deferred-frozen transfer.
Implantation rate | ≥ 35 weeks of gestation after the first single blastocyst embryo transfer according to fresh or deferred-frozen transfer.
  defined as the number of gestational sacs seen via transvaginal ultrasonography 4-5 weeks after embryo transfer, per number of embryos transferred
Cryopreservation thaw rate | ≥ 35 weeks of gestation after the first single blastocyst embryo transfer according to fresh or deferred-frozen transfer.
  defined as percentage of vitrified blastocysts which survive warming.
The incremental cost effectiveness ratio | ≥ 35 weeks of gestation after the first single blastocyst embryo transfer according to fresh or deferred-frozen transfer.
  using live birth rate as the effectiveness endpoint, after 35 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Khaled POCATE, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Cochin, Paris, France

REFERENCES:
- [Derived] Zaat T, Zagers M, Mol F, Goddijn M, van Wely M, Mastenbroek S. Fresh versus frozen embryo transfers in assisted reproduction. Cochrane Database Syst Rev. 2021 Feb 4;2(2):CD011184. doi: 10.1002/14651858.CD011184.pub3. PMID 33539543